CLINICAL TRIAL: NCT04705636
Title: Use of a Connected Companion in Children With Cystic Fibrosis - COMPANION-CF
Brief Title: Use of a Connected Companion in Children With Cystic Fibrosis
Acronym: COMPANION-CF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Saint-Brieuc (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHSB_202010_P3_COMPANION-CF; ID-RCB (Registry Identifier: 2020-A02971-38)
Record Dates: First submitted 2020-12-14; First posted 2021-01-12 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Cystic Fibrosis in Children; Chronic Disease
Keywords: Connected device; Long-term therapy; Pneumology; Adherence therapy; Pediatric research; Pediatric device support
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connected device (Experimental): Connected device for three months period to support children care
  Interventions: Device: Connected device named "Leo" from Ludocare society

INTERVENTIONS:
Device: Connected device named "Leo" from Ludocare society — Connected device named "Leo" from Ludocare society will be allocated to each child for three-months period. During this time, child will be helped to take all of his medication and specific care by this connected device.

SUMMARY:
The study will be conducted over a 6 months period. For the first three months, the child will be accompagned with a connected companion. After this period, the companion will be removed for three months in oder to prove this companion could improve treatment adherence for children suffering from cytolisis fibrosis.

This study will be conducted at the University Hospital Center of Rennes and Hospital Center of Saint-Brieuc.

DETAILED DESCRIPTION:
In developed countries, chronic diseases with long-term therapy adherence is about 50%, according to the WHO report, and the adherence rate for regular intake of preventive therapies decreases to 28%.

For cystic fibrosis, rates are not much higher. Optimistic articles report an average compliance rate of 60%. Other articles report a rate of 50% which varies according to the age of the patient, the intake treatment complexity and burdensome drug treatment (physiotherapy achieves the lowest adherence with 38%), the disease understanding and the interest of treatment persuasion. Low adherence can also be the result of incorrect use of administration devices, for example for inhaled treatments. Technical errors are very frequent and affect around 30% of patients.

Families with children suffering from cystic fibrosis need daily support. Health professionals need to relay their recommendations at home. This is why new and funny tools dedicated to children with chronic illnesses are needed.

This trial will study the impact of connected companion named LEO® created by Ludocare company.

Study will be conducted as :

* V0 : Companion given to the child
* V1 : Companion removed after 3 months of use
* V2 : Follow-up done between 1 and 3 months after the period without companion

ELIGIBILITY:
Inclusion Criteria:

* Child volunteer from 3 to 11 years old
* Affected by cystic fibrosis
* With a prescription containing at least two medications twice a day
* Affiliation to the national health insurance
* Child and holder of the exercise of parental authority understands and speaks French
* The person exercising parental authority must have reached the age of majority.
* Collection of the written consent of one of the holders of the exercise of parental authority

Exclusion Criteria:

* Non-voluntary child, under 3 years of age or over 12 years of age
* Family reluctant to technology
* Family without smartphone and/or wifi connection
* Failure to obtain the written consent of one of the holders of the exercise of parental authority
* Child involved in research involving the human person

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate therapeutic adherence of children with cystic fibrosis aged 3 to 11 years with help of a connected medical companion | Through study completion, up to 6 months
  The main evaluation criterion will be the overall compliance of the cohort in percentage terms. These data from connected companion will be refined for each type of treatment: pancreatic extracts, inhaled treatments, CFTR modulator, antibiotics, vitamins, laxative treatment, antacids, bile acids, food supplements, physiotherapy. For each treatment, the data "take" or "not take" will be treated by device and provide for statistical analysis in percentage. Each percentage will be grouped in global percentage will be therapeutic adherence all over study.

SECONDARY OUTCOMES:
Study of the reasons of low compliance or difficulties in taking the treatments | At the inclusion
  Questionnaire for parents with up to 15 treatments which provide the major difficulties (to be indicated in order, from the most difficult to the simplest, with checked answers; no specific scale available)
Assess the psycho-social impact of treatment and illness | At the inclusion
  Questionnaire for parents on child's behaviours in regard to taking treatment and illness (scale from 0 to 10, , highers scores mean better outcome)
Assess child's autonomy regarding his treatments | 3 months
  Reporting in connected device
Assess the intake treatments quality | At the inclusion
  Questionnaire for parents on difficulties frequency with checked answers (no specific scale available)
Evaluate any negative impacts associated with the use of the robot | 3 months
  Questionnaire for parents on difficulties linked to the use of the robot with scale from 0 to 10, highers scores mean better outcome, and open ended questions (no specific scale is available)
Evaluate any negative impacts associated with the use of the robot | 4 to 6 months
  Questionnaire for parents on difficulties linked to the use of the robot with scale from 0 to 10, highers scores mean better outcome, and open ended questions (no specific scale is available)
Assess the psycho-social impact of treatment and illness | at the inclusion
  Questionnaire for children on his relation to his illness and his treatments (Color gradient scale with expressive smiley : red (sad), orange (a little bit sad), yellow (neutral), light green (good), dark green (very good)
Assess the psycho-social impact of treatment and illness | 3 months
  Questionnaire for children on his relation to his illness and his treatments (Color gradient scale with expressive smiley : red (sad), orange (a little bit sad), yellow (neutral), light green (good), dark green(very good)
Assess the psycho-social impact of treatment and illness | 4 to 6 months
  Questionnaire for children on his relation to his illness and his treatments (Color gradient scale with expressive smiley : red (sad), orange (a little bit sad), yellow (neutral), light green (good), dark green(very good)
Study of the reasons of low compliance or difficulties in taking the treatments | 3 months
  Questionnaire for parents with up to 15 treatments which provide the major difficulties (to be indicated in order, from the most difficult to the simplest, with checked answers; no specific scale available)
Assess the psycho-social impact of treatment and illness | 3 months
  Questionnaire for parents on child's behaviours in regard to taking treatment and illness (scale from 0 to 10, , highers scores mean better outcome)
Assess the intake treatments quality | 3 months
  Questionnaire for parents on difficulties frequency with checked answers (no specific scale available)
Study of the reasons of low compliance or difficulties in taking the treatments | 4 to 6 months
  Questionnaire for parents with up to 15 treatments which provide the major difficulties (to be indicated in order, from the most difficult to the simplest, with checked answers; no specific scale available)
Assess the psycho-social impact of treatment and illness | 4 to 6 months
  Questionnaire for parents on child's behaviours in regard to taking treatment and illness (scale from 0 to 10, , highers scores mean better outcome)
Assess child's autonomy regarding his treatments | 4 to 6 months
  Reporting in connected device
Assess the intake treatments quality | 4 to 6 months
  Questionnaire for parents on difficulties frequency with checked answers (no specific scale available)

CONTACTS AND LOCATIONS:
Overall Officials: Marie JAMIN, Principal Investigator — Centre Hospitalier de Saint-Brieuc
Locations (2):
- France (2):
  - Chu Rennes, Rennes
  - Centre Hospitalier de Saint-Brieuc, Saint-Brieuc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De Geest S, Sabate E. Adherence to long-term therapies: evidence for action. Eur J Cardiovasc Nurs. 2003 Dec;2(4):323. doi: 10.1016/S1474-5151(03)00091-4. No abstract available. PMID 14667488
- [Result] Jentzsch NS, Camargos PAM, Colosimo EA, Bousquet J. Monitoring adherence to beclomethasone in asthmatic children and adolescents through four different methods. Allergy. 2009 Oct;64(10):1458-1462. doi: 10.1111/j.1398-9995.2009.02037.x. Epub 2009 Mar 28. PMID 19416142
- [Result] Zindani GN, Streetman DD, Streetman DS, Nasr SZ. Adherence to treatment in children and adolescent patients with cystic fibrosis. J Adolesc Health. 2006 Jan;38(1):13-7. doi: 10.1016/j.jadohealth.2004.09.013. PMID 16387243
- [Result] Conway SP, Pond MN, Hamnett T, Watson A. Compliance with treatment in adult patients with cystic fibrosis. Thorax. 1996 Jan;51(1):29-33. doi: 10.1136/thx.51.1.29. PMID 8658364
- [Result] Arias Llorente RP, Bousono Garcia C, Diaz Martin JJ. Treatment compliance in children and adults with cystic fibrosis. J Cyst Fibros. 2008 Sep;7(5):359-67. doi: 10.1016/j.jcf.2008.01.003. Epub 2008 Mar 4. PMID 18304896
- [Result] Sanchis J, Gich I, Pedersen S; Aerosol Drug Management Improvement Team (ADMIT). Systematic Review of Errors in Inhaler Use: Has Patient Technique Improved Over Time? Chest. 2016 Aug;150(2):394-406. doi: 10.1016/j.chest.2016.03.041. Epub 2016 Apr 7. PMID 27060726
- [Result] O'Donohoe R, Fullen BM. Adherence of subjects with cystic fibrosis to their home program: a systematic review. Respir Care. 2014 Nov;59(11):1731-46. doi: 10.4187/respcare.02990. Epub 2014 Jul 15. PMID 25233386
- [Result] Britto MT, Rohan JM, Dodds CM, Byczkowski TL. A Randomized Trial of User-Controlled Text Messaging to Improve Asthma Outcomes: A Pilot Study. Clin Pediatr (Phila). 2017 Dec;56(14):1336-1344. doi: 10.1177/0009922816684857. Epub 2017 Jan 5. PMID 28056541
- See also: Maladies : Comment les applications et objets connectés peuvent aider les enfants à prendre leur traitement ? — https://www.20minutes.fr/sante/2660383-20191129-maladies-comment-applications-objets-connectes-peuvent-aider-enfants-prendre-traitement